CLINICAL TRIAL: NCT04240704
Title: A Phase I/Ib Open-label, Multi-center Dose Escalation Study of JBH492 in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL) and Non-Hodgkin's Lymphoma (NHL)
Brief Title: Safety and Preliminary Efficacy of JBH492 Monotherapy in Patients With CLL and NHL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business, strategic, and development considerations and not due to any safety concerns
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CJBH492A12101; 2019-002666-12 (EudraCT Number)
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Non-Hodgkins Lymphoma; Chronic Lymphocytic Leukemia
Keywords: CLL; NHL; CCR7; JBH492; ADC; Chronic Lymphocytic Leukemia; Non-Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JBH492 single agent (Experimental): Patients with R/R CLL or NHL
  Interventions: Drug: JBH492

INTERVENTIONS:
Drug: JBH492 — Anti-CCR7 antibody-drug conjugate (ADC)

SUMMARY:
The purpose of the First-In-Human study was to assess the safety, tolerability, pharmacokinetics (PK), immunogenicity and preliminary efficacy of JBH492 as single agent.

DETAILED DESCRIPTION:
This was a FIH, open-label, phase I/Ib, multi-center study, which consisted of a dose escalation part of JBH492 as a single agent, followed by an expansion part. The escalation part was conducted in patients with relapsed/refractory chronic lymphocytic leukemia (r/r CLL) and Non-Hodgkin's Lymphoma (r/r NHL). Once the maximum tolerated dose/recommended dose (MTD/RD) of single agent JBH492 was determined, the study continued with an expansion part with single agent JBH492 in defined patient populations.

ELIGIBILITY:
Inclusion Criteria:

For patients with CLL:

• Confirmed diagnosis of chronic lymphocytic leukemia (CLL)

For patients with NHL:

* Histologically confirmed diagnosis of B- or T-cell non-Hodgkins lymphoma (NHL).
* Must have a site of disease amenable to biopsy, and be suitable and willing to undergo study required biopsies at screening and during therapy.

Exclusion Criteria, applicable to both CLL and NHL:

* History of anaphylactic or other severe hypersensitivity/infusion reactions to ADCs, monoclonal antibodies (mAbs) and/or their excipients such that the patient in unable to tolerate immunoglobulin/monoclonal antibody administration
* Any prior history of treatment with maytansine (DM1 or DM4)-based ADC
* Known intolerance to a maytansinoid
* Patients with any active or chronic corneal disorders
* Patients who have any other condition that precludes monitoring of the retina or fundus
* Patients with active CNS involvement are excluded, except if the CNS involvement has been effectively treated and provided that local treatment was completed >4 weeks before first dose of study treatment. Patients that have been effectively treated for CNS disease and are stable under systemic therapy may be enrolled provided all other inclusion and exclusion criteria are met. Patients who received prophylactic intrathecal treatment are eligible, if treatment discontinued >5 half-lives prior to the first dose of study treatment
* Impaired cardiac function or clinically significant cardiac disease
* Known history of Human Immunodeficiency Virus (HIV) infection
* Active HBV or HCV infection. Patients whose disease is controlled under antiviral therapy should not be excluded. Patients who are anti-HBcAb positive should be HBsAg negative and HBV-DNA negative to be eligible

Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of dose limiting toxicities (DLTs) | 32 months
  A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value that occurs during the first cycle of treatment with JBH492 and meets any of the protocol specified criteria, unless incontrovertibly related to underlying disease, intercurrent illness or concomitant medications.
Incidence and severity of Adverse Events (AEs) | 32 months
  An adverse event ( treatment emergent) is defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) that occur after patient's signed informed consent has been obtained.
Incidence and severity of Serious Adverse Events (SAEs) | 32 months
  A Serious adverse event (SAE) is defined as one of the following:
  * Is fatal or life-threatening
  * Results in persistent or significant disability/incapacity
  * Constitutes a congenital anomaly/birth defect
  * Is medically significant
  * Requires inpatient hospitalization or prolongation of existing hospitalization.
Number of patients with dose interruptions | 32 months
  Tolerability measured by the number of subjects who have interruptions of study treatment and reason for interruptions
Number of patients with dose reductions | 32 months
  Tolerability measured by the number of subjects who have reductions of study treatment and reason for reductions
Dose intensity | 32 months
  Tolerability measured by the dose intensity of study drug, Relative Dose intensity for subjects with non-zero duration of exposure is computed as the ratio of dose intensity and planned dose intensity

SECONDARY OUTCOMES:
Overall response rate (ORR) | 32 months
  The overall response rate (ORR), defined as the proportion of subjects with best overall response (BOR) of complete response (CR) or partial response (PR), as per local review and according to the iwCLL guideline (CLL) or Lugano Classification (NHL).
Best overall response (BOR) | 32 months
  The best overall response (BOR) is the best reponse recorded in a patient from the start of treatment until disease progression.
Duration of Response (DOR) | 32 months
  The time between the date of first documented response (CR or PR) and the date of first documented progression or death due to underlying cancer.
Progression Free Survival (PFS) | 32 months
  PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause
Pharmacokinetics (PK) parameter AUClast | 32 months
  The area under the plasma concentration-time curve (AUC) of JBH492 from time zero to the last measurable concentration sampling time (tlast) for four analytes (total antibody, total antibody-drug-conjugate, DM4, sDM4)
PK parameter AUCinf | 32 months
  The AUC from time zero to infinity (mass × time × volume-1) for four analytes (total antibody, total antibody-drug-conjugate, DM4, sDM4)
PK parameter AUCtau | 32 months
  The AUC calculated to the end of a dosing interval (tau) (mass × time × volume-1) for four analytes (total antibody, total antibody-drug-conjugate, DM4, sDM4)
PK parameter Cmax and Cmin | 32 months
  The maximum (peak) and minimum observed serum drug concentration (mass × volume-1) for four analytes (total antibody, total antibody-drug-conjugate, DM4, sDM4)
PK parameter Tmax | 32 months
  The time to reach maximum (peak) serum drug concentration (time) for four analytes (total antibody, total antibody-drug-conjugate, DM4, sDM4)
PK parameter T1/2 | 32 months
  The elimination half-life associated with the terminal slope (λz) of a semi logarithmic concentration-time curve (time) for four analytes (total antibody, total antibody-drug-conjugate, DM4, sDM4)
Incidence of anti-JBH492 antibodies | 32 months
  Number of subjects with anti-JBH492 antibodies (Anti-Drug Antibodies)

CONTACTS AND LOCATIONS:
Locations (8):
- Novartis Investigative Site, Helsinki, Finland
- Germany (2):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Freiburg im Breisgau
- Novartis Investigative Site, Tel Aviv, Israel
- Novartis Investigative Site, Chuo Ku, Tokyo, Japan
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18330
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2738